CLINICAL TRIAL: NCT01686503
Title: Comparison of the Immunogenicity of Various Inactivated Polio Vaccine Booster Doses by Intradermal vs. Intramuscular Routes in HIV-Infected Subjects
Brief Title: Intradermal Versus Intramuscular Polio Vaccine Booster in HIV-Infected Subjects
Acronym: IDIPV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: NanoPass Technologies Ltd (Industry)
Responsible Party: Principal Investigator, Stephanie Troy, Assistant Professor, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Doris Duke CF-2012061
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-01

CONDITIONS: Polio Immunity
MeSH Terms: interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2/5 dose intradermal IPV (Experimental): Participants in this arm will receive 2/5 dose (0.2 mL) of inactivated polio vaccine (IPOL, Sanofi Pasteur) as a one-time dose intradermally using the NanoPass MicronJet 600 microneedle device
  Interventions: Drug: IPOL (Sanofi Pasteur) inactivated polio vaccine booster dose
- 1/5 dose intradermal IPV (Experimental): Participants in this study arm will receive 1/5 dose (0.1 mL) of inactivated polio vaccine (IPOL, Sanofi Pasteur) as a one time dose intradermally using the NanoPass MicronJet 600 microneedle device.
  Interventions: Drug: IPOL (Sanofi Pasteur) inactivated polio vaccine booster dose
- full dose intramuscular IPV (Active Comparator): Participants in this study arm will receive the standard full dose (0.5 mL) of inactivated polio vaccine (IPOL, Sanofi Pasteur) as a one time dose intramuscularly.
  Interventions: Drug: IPOL (Sanofi Pasteur) inactivated polio vaccine booster dose
- 2/5 dose intramuscular IPV (Active Comparator): Participants in this study arm will receive 2/5 dose (0.2 mL) inactivated polio vaccine (IPOL, Sanofi Pasteur) as a one time dose intramuscularly.
  Interventions: Drug: IPOL (Sanofi Pasteur) inactivated polio vaccine booster dose

INTERVENTIONS:
Drug: IPOL (Sanofi Pasteur) inactivated polio vaccine booster dose — Depending on study arm, participants will receive 0.2 mL intradermally, 0.1 mL intradermally, 0.5 mL intramuscularly, or 0.2 mL intramuscularly.
  Other Names: IPOL (Sanofi Pasteur)

SUMMARY:
The purpose of this study is to determine whether a lower dose of inactivated polio vaccine (IPV) injected into the skin (intradermal administration) can work equally well or better than the standard dose injected into the muscle (intramuscular administration). There are more immune cells in the skin than in the muscle, and other vaccines have been shown to require a lower dose when administered intradermally. The study is being done in participants infected with HIV because HIV-infected people are known to respond less well to vaccines than other groups, so it is particularly important to know if IPV might work better in HIV-infected people if administered intradermally.

If it is possible to lower the dose of IPV by intradermal administration, this would make inactivated polio vaccine more affordable in the developing countries where it is most needed

DETAILED DESCRIPTION:
Oral polio vaccine (OPV) will not be sufficient to eradicate polio. OPV has failed to provide adequate polio immunity in certain immunocompromised populations, such as people with AIDS. Also, OPV can mutate and form neurovirulent strains capable of causing polio outbreaks. Inactivated polio vaccine (IPV), which cannot mutate into neurovirulent strains and which is more effective in populations that have failed to respond to OPV, will be needed globally to eradicate polio, but it is unaffordable for many developing countries. Because there are more immune cells in the skin than in the muscle, intradermal administration of IPV may be a way to increase the efficacy and reduce the dose (and thus the cost) of IPV. We plan to conduct a clinical trial randomizing 231 HIV-infected adults to receive a booster of two-fifths dose intradermal IPV, one-fifth dose intradermal IPV, full dose intramuscular IPV, or two-fifths dose intramuscular IPV. We will measure polio immunity before and after vaccine administration. Through this study, we will determine the optimal booster dose of intradermal IPV, whether intradermal works better than intramuscular IPV administration, and whether intradermal IPV is effective in an immunocompromised population. The data from this trial could contribute to global polio eradication.

ELIGIBILITY:
Inclusion Criteria:

* documented HIV infection
* age of at least 18 years old
* HIV viral load <400 on the most recent test

Exclusion Criteria:

* current acute moderate to severe illness (demonstrated by fever over 100.4 Fahrenheit, shortness of breath, altered mental status, or by judgment of the primary clinician)
* current pregnancy
* history of allergic reaction to a polio shot,
* history of a life-threatening allergic reaction to neomycin, streptomycin, or polymyxin B

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Troy, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- C3ID Clinic, Eastern Virginia Medical School, Norfolk, Virginia, United States

REFERENCES:
- [Result] Troy SB, Kouiavskaia D, Siik J, Kochba E, Beydoun H, Mirochnitchenko O, Levin Y, Khardori N, Chumakov K, Maldonado Y. Comparison of the Immunogenicity of Various Booster Doses of Inactivated Polio Vaccine Delivered Intradermally Versus Intramuscularly to HIV-Infected Adults. J Infect Dis. 2015 Jun 15;211(12):1969-76. doi: 10.1093/infdis/jiu841. Epub 2015 Jan 7. PMID 25567841

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/5 Dose Intadermal IPV: Participants in this study arm will receive 1/5 dose (0.1 mL) of inactivated polio vaccine (IPOL, Sanofi Pasteur) as a one time dose intradermally using the NanoPass MicronJet 600 microneedle device.
  IPOL (Sanofi Pasteur) inactivated polio vaccine booster dose: Depending on study arm, participants will receive 0.2 mL intradermally, 0.1 mL intradermally, 0.5 mL intramuscularly, or 0.2 mL intramuscularly.
Period: Overall Study
Arm/Group | 2/5 Dose Intradermal IPV | 1/5 Dose Intadermal IPV | Full Dose Intramuscular IPV | 2/5 Dose Intramuscular IPV
Started | 66 | 66 | 66 | 33
Completed | 65 | 63 | 64 | 32
Not Completed | 1 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2/5 Dose Intradermal IPV | 1/5 Dose Intadermal IPV | Full Dose Intramuscular IPV | 2/5 Dose Intramuscular IPV | Total
Number analyzed (Participants) | 66 | 66 | 66 | 33 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10) | 45 (11) | 46 (11) | 46 (11) | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 21 | 7 | 76
  Male | 42 | 42 | 45 | 26 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 0 | 0 | 8
  Not Hispanic or Latino | 62 | 60 | 66 | 33 | 221
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 47 | 48 | 47 | 21 | 163
  White | 19 | 17 | 19 | 11 | 66
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Most recent CD4 count [Mean (Standard Deviation); unit: cells/mm^3] | 669 (361) | 630 (331) | 676 (354) | 569 (260) | 645 (338)
Currently on antiretroviral therapy [Number; unit: participants] | 64 | 64 | 66 | 33 | 227
Diagnosis of AIDS in the record [Number; unit: participants] | 38 | 33 | 39 | 17 | 127
Year diagnosed with HIV [Mean (Standard Deviation); unit: calendar year] | 2001 (8) | 2002 (8) | 2001 (8) | 2001 (9) | 2002 (8)
Born in the United States [Number; unit: participants] | 65 | 63 | 60 | 31 | 219
Lived or traveled internationally [Number; unit: participants] | 18 | 19 | 29 | 12 | 78
Reported receiving all childhood vaccines [Number; unit: participants] | 64 | 64 | 60 | 31 | 219
Current smoker [Number; unit: participants] | 38 | 31 | 23 | 13 | 105
Coinfected with hepatitis C [Number; unit: participants] | 12 | 10 | 6 | 5 | 33
Coinfected with hepatitis B [Number; unit: participants] | 7 | 4 | 2 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Post Booster Polio Neutralizing Antibody Titers
Description: Blood will be drawn at baseline and 4-6 weeks after receiving the vaccine booster dose. It will be spun down, and the serum frozen and stored at -80 degrees celsius. After all the participants have completed the study, all of the serum will be tested for polio neutralizing antibody titers.
Time Frame: 4-6 weeks after receiving the vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titers
Arm/Group | 2/5 Dose Intradermal IPV | 1/5 Dose Intadermal IPV | Full Dose Intramuscular IPV | 2/5 Dose Intramuscular IPV
Number analyzed (Participants) | 65 | 63 | 64 | 32
antibody titers
  Serotype 1 | 1715 [1174 to 2504] | 976 [730 to 1304] | 1249 [916 to 1705] | 1328 [795 to 2219]
  Serotype 2 | 2188 [1507 to 3178] | 1438 [984 to 2101] | 1489 [1041 to 2128] | 1938 [1232 to 3047]
  Serotype 3 | 2375 [1423 to 3963] | 1698 [1114 to 2588] | 1792 [1133 to 2835] | 2075 [1225 to 3514]

2. Secondary Outcome: Baseline Polio Neutralizing Antibody Titers
Description: serum polio neutralizing antibody titers prior to the vaccine booster
Time Frame: first visit
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titers
Arm/Group | 2/5 Dose Intradermal IPV | 1/5 Dose Intadermal IPV | Full Dose Intramuscular IPV | 2/5 Dose Intramuscular IPV
Number analyzed (Participants) | 65 | 63 | 64 | 32
antibody titers
  Serotype 1 | 44 [31 to 64] | 42 [29 to 59] | 42 [30 to 58] | 34 [20 to 56]
  Serotype 2 | 33 [24 to 44] | 53 [37 to 76] | 36 [26 to 51] | 44 [29 to 66]
  Serotype 3 | 14 [10 to 20] | 20 [14 to 28] | 16 [11 to 21] | 11 [7 to 16]

ADVERSE EVENTS:
Arm/Group | 2/5 Dose Intradermal IPV | 1/5 Dose Intadermal IPV | Full Dose Intramuscular IPV | 2/5 Dose Intramuscular IPV
Serious Adverse Events (participants affected / at risk) | 1/66 | 0/66 | 0/66 | 0/33
Other Adverse Events (participants affected / at risk) | 33/66 | 29/66 | 18/66 | 10/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2/5 Dose Intradermal IPV (N=66) | 1/5 Dose Intadermal IPV (N=66) | Full Dose Intramuscular IPV (N=66) | 2/5 Dose Intramuscular IPV (N=33)
Hospitalization for electrolyte imbalances secondary to alcohol withdrawal (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Occured one month after receiving the vaccine
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2/5 Dose Intradermal IPV (N=66) | 1/5 Dose Intadermal IPV (N=66) | Full Dose Intramuscular IPV (N=66) | 2/5 Dose Intramuscular IPV (N=33)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Redness at Injection Site (Skin and subcutaneous tissue disorders) | 19 (19) | 22 (22) | 4 (4) | 3 (3)
Swelling at Injection Site (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7) | 3 (3) | 2 (2)
Tenderness at Injection Site (General disorders) | 10 (10) | 8 (8) | 11 (11) | 5 (5)
Itching at injection site (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Higher baseline antibody titers than expected making it more difficult to detect differences between the study groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No